CLINICAL TRIAL: NCT02531178
Title: A Randomized, Double-Blind, Placebo-Controlled Study in Subjects With Rheumatoid Arthritis to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of ABBV-257
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Subcutaneous Injections of ABBV-257 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: M14-439; 2015-000094-12 (EudraCT Number)
Record Dates: First submitted 2015-07-14; First posted 2015-08-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- low dose ABBV-257 (Experimental): Low dose every other week (eow), Weeks 0-8
  Interventions: Biological: ABBV-257; Biological: Placebo
- Medium dose of ABBV-257 (Experimental): Medium dose every other week (eow), Weeks 0-8
  Interventions: Biological: ABBV-257; Biological: Placebo
- high dose of ABBV-257 (Experimental): high dose every other week (eow), Weeks 0-8
  Interventions: Biological: ABBV-257; Biological: Placebo

INTERVENTIONS:
Biological: ABBV-257 — subcutaneous injection
Biological: Placebo — Placebo for ABBV-257

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, multiple dose study designed to assess the safety, tolerability, pharmacokinetics, and immunogenicity of different dose levels of ABBV-257 given with methotrexate. ABBV-257 or placebo will be administered once every other week (EOW) for a total of 4 doses. Subjects will continue on their stable dose of methotrexate weekly throughout participation in the study.

This study will be conducted in approximately 24 subjects in 3 dose groups, with 8 subjects per group. Within each group, 6 subjects will be randomized to receive ABBV-257 and 2 subjects will receive placebo. Subjects participating in one dose group will be ineligible to participate in another dose group in the study.

DETAILED DESCRIPTION:
Multiple dose study designed to assess the safety, tolerability, pharmacokinetics, and immunogenicity of different dose levels of ABBV-257 given with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis based on the 2010 American College of Rheumatology (ACR)/European League against Rheumatism (EULAR) criteria, or ACR 1987 for patients with diagnosis prior 2011 ≥ 3 months.
* Except for methotrexate (MTX), the subject must have discontinued all disease modifying anti-rheumatic drugs (DMARD) for at least 5 half-lives before the first dose of study drug, and undergone cholestyramine washout if received Leflunomide within the past 3 months.
* Subject must have been on MTX therapy > 3 months and on a stable dose (7.5 - 25 mg/week), for at least 4 weeks prior to the first dose of study drug. Subject must be able to continue on stable dose of MTX for the duration of study participation.
* Body Mass Index (BMI) is 19 to 35, inclusive. (BMI is calculated as weight [kg] divided by height [m2].)
* Judged to be in good general health as determined by the Investigator based upon the results of medical history, laboratory profile, physical examination and 12-lead electrocardiogram (ECG) performed at screening

Exclusion Criteria:

* Evidence of anti-ABBV-257 antibody results in a pre-study serum sample.
* History of significant allergic reaction or significant sensitivity to any constituents of the study drug; or history of anaphylactic reaction to any agent (e.g., food products and bee sting); or history of a major reaction to any Immunoglobulin G (IgG) containing product.
* History of persistent chronic or active infection(s) requiring hospitalization or treatment with intravenous or oral antimicrobials/antibiotics within 30 days prior to initial study drug administration.
* History or evidence of active tuberculosis (TB) or the subject has evidence of risk factor for latent TB.
* Clinically significant abnormal screening laboratory results as evaluated by the Investigator, including serum values of Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) greater than 2.25 × the upper limit of normal, or creatinine greater than 1.5 × the upper limit of normal, or absolute neutrophil count < 1500 μ/L.
* Subject has any medical condition or illness other than RA that is not well controlled with treatment that would, in the opinion of the investigator, preclude study participation or interfere with other symptoms of Rheumatoid Arthritis (RA).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with adverse events | Up to day 193
  This will be collected through out the study
Change in Vital signs | From day 1 to day 193
  Vital signs including blood pressure and heart rate will be assessed
Change in Physical examination | From day 1 to day 193
  Changes in any physical exam assessed by the physician will be assessed.
Changes in Electrocardiogram (ECG) | From day 1 to day 193
  ECG measurements will be assessed
Maximum observed serum concentration (Cmax) | Up to day 50
  This will be assessed using non-compartmental methods.
Time to maximum observed serum concentration (Tmax) | Up to day 50
  This will be assessed using non-compartmental methods.

SECONDARY OUTCOMES:
Immunogenicity by measurement of Anti-drug antibody | Up to day 193
  Immunogenicity will be measured to see if the body has produced an immune response to ABBV-257

OTHER OUTCOMES:
American College of Rheumatology (ACR) 20 response rate | Up to day 193
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
American College of Rheumatology (ACR) 50 response rate | Up to day 193
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
American College of Rheumatology (ACR) 70 response rate | Up to day 193
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
Change in Disease Activity Score 28 | From day 1 to day 193
  Calculated from tender joint, swollen joint and high sensitive C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Mansikka, PhD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 139394, Berlin, Germany